CLINICAL TRIAL: NCT06614842
Title: Common Factors Group Psychotherapy for General Mental Health Concerns
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Inability for consistent recruitment.
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Nicholas C. Borgogna, Assistant Professor, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-300013539
Record Dates: First submitted 2024-09-24; First posted 2024-09-26 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Major Depression; Generalized Anxiety; Stress Disorder, Post Traumatic; Stress; Mental Disorders
Keywords: common factors psychotherapy
MeSH Terms: conditions — Depressive Disorder, Major; Generalized Anxiety Disorder; Stress Disorders, Post-Traumatic; Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Common Factors Group Therapy (Experimental): We will use a general common factors psychotherapy utilizing only psychotherapeutic techniques common to most forms of psychotherapy (e.g., listening and communication skills)
  Interventions: Behavioral: Common Factors Group Psychotherapy

INTERVENTIONS:
Behavioral: Common Factors Group Psychotherapy — This intervention will not contain active ingredients from established specific forms of psychotherapy (e.g., cognitive-behavioral therapy, dialectical behavioral therapy)

SUMMARY:
The current research will investigate the impact of general psychotherapy using common factors (i.e., techniques and communication skills that are common to all major forms of psychotherapy) to investigate whether mental health professionals can treat a variety of mental health concerns utilizing this general form of psychotherapy as opposed to specific forms of psychotherapy that may require specific trainings or education.

DETAILED DESCRIPTION:
The current research will investigate the impact of general psychotherapy using common factors (i.e., techniques and communication skills that are common to all major forms of psychotherapy) to investigate whether mental health professionals can treat a variety of mental health concerns utilizing this general form of psychotherapy as opposed to specific forms of psychotherapy that may require specific trainings or education.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Experiencing self-reported psychological distress

Exclusion Criteria:

* has engaged in self-harm within the last three months
* has attempted suicide within the last year
* has had an active plan to attempt suicide within the last 30 days
* currently diagnosed with any eating disorder
* has experienced hallucinations or delusions within the last 30 days
* has used narcotics within the last 7 days (heroin, meth, crack cocaine, opioids)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-01-17 (Actual); Primary Completion 2025-12-30 (Actual); Study Completion 2025-12-30 (Actual)

PRIMARY OUTCOMES:
Generalized Anxiety Disorder-7 Screener | At enrollment and at the end of treatment at 6 weeks
  Measure of anxiety symptoms. High scores more symptoms.
Patient Health Questionnaire-9 Screener | At enrollment and at the end of treatment at 6 weeks
  Measure of depressive symptoms. High scores more symptoms.
Patient Checklist-5 | At enrollment and at the end of treatment at 6 weeks
  Measure of post-traumatic stress symptoms. High scores more symptoms.
Yale-Brown Obsessive Compulsive Scale | At enrollment and at the end of treatment at 6 weeks
  Measure of obsessive compulsive disorder symptoms. High scores more symptoms.
Alcohol Use Disorders Identification Test | At enrollment and at the end of treatment at 6 weeks
  Measure of concerning alcohol use. High scores more symptoms.
National Institute of Drug Abuse Modified Alcohol, Smoking, and Substance Involvement Screening Test | At enrollment and at the end of treatment at 6 weeks
  Measure of substance use. High scores more use.

SECONDARY OUTCOMES:
Life Quality Scale | At enrollment and at the end of treatment at 6 weeks
  Measure of life quality. High scores better life quality.
Experiential Avoidance Rating Scale | At enrollment and at the end of treatment at 6 weeks
  Measure of experiential avoidance. High scores more symptoms.

OTHER OUTCOMES:
Therapeutic Alliance Scale | At conclusion of therapy after 6 weeks.
  Measure of patient-therapist alliance during therapy. High scores better alliance.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Borgogna, PhD, Principal Investigator — University of Alabama at Birmingham; Drew Whittington, MS, MA, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Yes
All de-identified data collected will be available2
Time Frame: When results are published
Access Criteria: Requesting researchers